CLINICAL TRIAL: NCT06391671
Title: The Stress-obesity Axis: a Metabolomics Approach Towards Personalized Nutrition in Adolescents (FAME)
Brief Title: The Stress-obesity Axis: a Metabolomics Approach Towards Personalized Nutrition in Adolescents
Acronym: FAME
Status: Recruiting | Type: Observational
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: BC-10583
Record Dates: First submitted 2024-04-19; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Pediatric Obesity
Keywords: Metabolomic; Mass spectrometry
MeSH Terms: conditions — Pediatric Obesity | interventions — Defecation; Surveys and Questionnaires; Demography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples With DNA — Stool, saliva and hair
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Overweight/obese: BMI-Z > 25
  Interventions: Other: Collection of anthropometric data, biological samples (stool, saliva and hair), questionnaires (demographic data, psychological data, medical data)
- Normal weight: BMI-Z < 25
  Interventions: Other: Collection of anthropometric data, biological samples (stool, saliva and hair), questionnaires (demographic data, psychological data, medical data)

INTERVENTIONS:
Other: Collection of anthropometric data, biological samples (stool, saliva and hair), questionnaires (demographic data, psychological data, medical data) — Saliva and feces are collected at the families home. A questionnaire is filled in by the participant (psychological) and parents (demographical and medical info). Upon consultation we are collecting anthropometric data (date of birth, length, weight, abdominal circumference, Tanner pubertal stage, etc.)

SUMMARY:
The ultimate aim of this project is to establish a validated strategy that allows for personalized intervention in adolescents (11 to 17 years) whom are assigned a state of overweight or obesity.

The investigators will assess the following hypotheses:

* Weight condition is reflected by the fecal metabolome (WP1)
* Emotional stress is implicated in weight condition (WP1)
* Functionality of the gut microbiome is related to the diet-stress-obesity axis (WP2)
* Dietary pattern impacts the fecal metabolome and gut microbiome (WP2)
* Personalized dietary intervention outperforms generalized dietary approaches (WP3)

Participants will:

* Produce a saliva, stool and hair sample
* Fill in questionnaires regarding mental health, medical health and demographic information
* Fill in a food frequency questionnaire and a 24-hrecalls
* Be measured (height, weight, fat% and waist circumference)

The samples will be analyzed using a technique called metabolomics to identify biomarker candidates with diagnostic and/or prognostic potential. Additionally, microbiome analysis will be performed to map the microbiome of all groups.

DETAILED DESCRIPTION:
In WP1, the investigators will assess the metabolic mechanisms underlying the obesity pathology in adolescents, whereby the involvement of emotional stress, will be of particular interest. To this end, a dual strategy fecal metabolomics will be performed: targeted profiling and untargeted fingerprinting. A major objective in this respect is to metabolically segregate between the overweight/obesity and normal weight condition as well as to reveal metabolic singularities that specifically relate to emotional stress. Fecal material, saliva and a hair sample will be collected from adolescents (11 to 17 years). Assignment of a participant's stress state will be performed post-hoc and based on hair cortisol concentrations and scores from the psychological questionnaires. The samples will be collected at home and have to be frozen immediately after sample collection. The samples will be analyzed using a technique called metabolomics, using UHPLC-HRMS (Ultra-High Performance Liquid Chromatography coupled to High-Resolution Mass Spectrometry).

In WP2 the investigators will assess the microbiome and diet as drivers for obesity. Fecal samples will be subjected to DNA extraction and whole-metagenome shotgun sequencing will be performed using the Illumina HiSeq 2500 system (151 bp paired-end reads; Novogene). In order to collect data about both long- and short-term dietary intakes, participants will be provided with a FFQ and a 24-h recall.

Eventually, discovery of metabolite marker signatures and elucidation of mechanistic pathways will offer opportunities to stratify obese adolescents according to emotional stress status, microbial composition and dietary preferences.

In WP3, the new data from WP1/2 will be translated in personalized dietary recommendations. The investigators will assess the potential of dietary interventions focused on nutrient quality (not energy-reduced) to affect the stress-obesity axis directly or by gut microbial modulation. After ethical approval, the dietary intervention study will include up to 20 individuals that were allocated to the overweight/obesity group. In our 3-month personalized intervention, separate menus for each participant will be prepared by our dietician. Based on WP1/2 and literature evidence, appropriate changes in nutrients will be aimed for. At different points in time, fecal samples will be collected, aliquoted and biobanked at -80°C. Fecal samples will be used for polar metabolomics and lipidomics analyses and microbiome metasequencing. At the start and after the 3-months intervention, fasting blood samples will be taken for clinical biomarkers (glucose, insulin, cholesterol, cytokines, ...). In addition, indirect calorimetry will determine resting energy expenditure. Anthropometric measures include BMI, waist and fat%. Questionnaires cover emotional eating (DEBQ), satiety, physical activity, sleep and quality-of-life (KINDL). Study volunteers will be asked to fill out an FFQ and 3-day 24-h recall to assess dietary habits prior to the trial.

ELIGIBILITY:
Inclusion Criteria:

* Age 11-17 years

Exclusion Criteria:

* Obesity/overweight
* Type 1 diabetes
* Medical conditions including pancreatic failure
* Developmental and hormonal disorders. E.g. thyroid problems, adrenal problems, Kallmann's syndrome, Klinefelter's syndrome, Prader-Willi syndrome (PWS), Congenital hypogonadotropic hypogonadism (CHH), ...
* Pregnancy
* In treatment with systemic concentrations of corticosteroids (cortisone). Eg cortisone/betamethasone/Dexamethasone/Fludrocortisone/Hydrocortisone in pill form or administration by injections.

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Volunteers with normall weight and overweight/obesity are being recruited from several hospitals (UZ Ghent, AZ Jan Palfijn, UZ Antwerpen, ZNA Middelheim, AZ Delta Roeselare, UZ Brussel, UZ Leuven, Onze-Lieve-Vrouw Ziekenhuis Aalst, AZ Sint-Lucas Brugge, AZ Sint-Elizabeth Zottegem, Zeepreventorium, Clairs Vallons) and schools (Don-Bosco Sint-Denijs-Westrem, Leiepoort Deinze, Broederschool Sint-Niklaas, SFI Melle) in Belgium
Sampling Method: Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2022-01-11 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Metabolomics | Samples will be analyzed in the 4th quarter of 2024.
  Saliva and fecal samples will be analyzed using a technique called metabolomics, which analyses all small molecules (metabolites) present in a biological fluid. These metabolites will be used to find biomarkers that are related to the disease and could have diagnostic or prognostic potential. Additionally, these metabolites could give more insights into the development and maintenance of the disease.

SECONDARY OUTCOMES:
Microbiome analysis | Microbiome analyses will be performed at the start of 2025
  The microbiomes of all groups will be analyzed because it has been described in literature that the microbiome can differ between healthy and obese individuals
Stress levels | Hair cortisol analyses will be conducted in the first quarter of 2025. Data processing of the questionnaires is an ongoing process, to be completed by the last quarter of 2024
  Assignment of a participant's stress state will be performed based on hair cortisol concentrations, and scores from the Perceived Stress Scale (PSS), the Children's Depression Inventory 2 (CDI-2) and the Rosenberg Self-Esteem Scale (RSES) questionnaires. A summary chronic stress variable will be calculated by adding up the four z-score-transformed variables to give them equal weight
Food frequency questionnaire | FFQ data are being analyzed continuously and will be finished when the sample collection is finished (estimated by the end of 2024)
  To collect data about dietary intakes, participants are provided with an FFQ. Participants are required to indicate the frequency of consumption for each food of interest, ranging from (almost) never, to a few times a week, (almost) daily, to multiple times a day. All responses are encoded into numerical values, representing the frequency of consumption for specific foods.

CONTACTS AND LOCATIONS:
Overall Officials: Stefaan de Henauw, Prof, Principal Investigator — University Hospital, Ghent
Locations (7):
- Belgium (7):
  - AZ Jan Palfijn Gent, Oost-Vlaanderen, Belgium, 9000, Ghent, Oost-Vlaanderen
  - Ghent University Hospital, Ghent, Oost-Vlaanderen
  - Clairs Vallons, Ottignies-Louvain-la-Neuve, Waals Brabant
  - Zeepreventorium, De Haan, West-Vlaanderen
  - AZ Delta, Roeselare, West-Vlaanderen
  - UZ Antwerpen, Antwerp
  - ZNA Middelheim, Antwerp

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researchers